CLINICAL TRIAL: NCT03161093
Title: A Phase 3 Randomized, Double-blind, Multi-dose, Placebo and Naproxen-Controlled Study to Evaluate the Efficacy and Safety of Fasinumab in Patients With Pain Due to Osteoarthritis of the Knee or Hip
Brief Title: A Study to Determine the Safety and the Efficacy of Fasinumab Compared to Placebo and Naproxen for Treatment of Adults With Pain From Osteoarthritis of the Knee or Hip
Acronym: FACT OA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R475-OA-1611; 2016-005020-29 (EudraCT Number)
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — fasinumab; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fasinumab dosing regimen 1 (Experimental): Fasinumab Subcutaneous (SC) dosing regimen 1 and naproxen-matching placebo oral
  Interventions: Drug: Fasinumab; Drug: Naproxen-matching placebo
- Fasinumab dosing regimen 2 (Experimental): Fasinumab SC dosing regimen 2 and naproxen-matching placebo oral
  Interventions: Drug: Fasinumab; Drug: Naproxen-matching placebo
- Fasinumab-matching placebo and naproxen (Experimental)
  Interventions: Drug: Naproxen; Drug: Fasinumab-matching placebo
- Fasinumab-matching placebo and naproxen-matching placebo (Experimental)
  Interventions: Drug: Fasinumab-matching placebo; Drug: Naproxen-matching placebo

INTERVENTIONS:
Drug: Fasinumab — Solution for injection in pre-filled syringe
  Other Names: REGN475
  Arms: Fasinumab dosing regimen 1; Fasinumab dosing regimen 2
Drug: Naproxen — Pharmaceutical form: Capsule
  Arms: Fasinumab-matching placebo and naproxen
Drug: Fasinumab-matching placebo — Solution for injection in pre-filled syringe
  Arms: Fasinumab-matching placebo and naproxen; Fasinumab-matching placebo and naproxen-matching placebo
Drug: Naproxen-matching placebo — Capsule
  Arms: Fasinumab dosing regimen 1; Fasinumab dosing regimen 2; Fasinumab-matching placebo and naproxen-matching placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of fasinumab compared with placebo, when administered for up to 16 weeks in patients with pain due to osteoarthritis (OA) of the knee or hip.

The secondary objectives of the study are:

1. To evaluate the efficacy of fasinumab compared with naproxen, when administered for up to 16 weeks in patients with pain due to OA of the knee or hip
2. To evaluate the efficacy of fasinumab compared with placebo, when administered for up to 44 weeks in patients with pain due to OA of the knee or hip
3. To assess the safety and tolerability of fasinumab compared with naproxen, when administered for up to 16 weeks in patients with pain due to OA of the knee or hip
4. To assess the safety and tolerability of fasinumab compared with naproxen, when administered for up to 52 weeks in patients with pain due to OA of the knee or hip
5. To assess the safety and tolerability of fasinumab compared with naproxen, when administered for up to 104 weeks in patients with pain due to OA of the knee or hip
6. To evaluate the pharmacokinetic (PK) profile of fasinumab administered to patients with pain due to OA of the knee or hip for up to 52 weeks
7. To evaluate the PK profile of fasimumab administered to patients with pain due to OA of the knee or hip for up to 104 weeks
8. To evaluate the immunogenicity of fasinumab administered to patients with pain due to OA of the knee or hip for up to 52 weeks
9. To evaluate the immunogenicity of fasinumab administered to patients with pain due to OA of the knee or hip for up to 104 weeks
10. To evaluate the efficacy of fasinumab compared with naproxen, when administered for up to 44 weeks in patients with pain due to OA of the knee or hip

ELIGIBILITY:
Inclusion Criteria include, but are not limited to, the following:

Year 1:

1. Male and female patients, at least 18 years of age, at screening
2. A clinical diagnosis of OA of the knee or hip based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2 for the index joint) at the screening visit
3. Moderate to severe pain in the index joint defined at both the screening and randomization visits
4. Willing to discontinue current pain medications and to adhere to study requirements for rescue treatments (acetaminophen/paracetamol) to be taken as needed with a maximum daily dose of 2500 mg (countries where 500 mg strength tablets/capsules are available) or 2600 mg (countries where 325 mg strength tablets/capsules are available)
5. A history of at least 12 weeks of analgesics use for pain due to OA of the knee or hip, as defined by:

   1. Inadequate pain relief from acetaminophen/paracetamol AND
   2. Intolerance to or inadequate pain relief from opioid or tramadol therapy, unwillingness to take opioid or tramadol therapy for a medically acceptable reason, or lack of access to an opioid or to tramadol
6. Currently using a stable dose of NSAID.
7. Willing to discontinue glucosamine sulfate and chondroitin sulfate treatments during the initial 16 weeks of treatment
8. Stable treatment with glucosamine sulfate and chondroitin sulfate treatments must be stopped during the pre-randomization period
9. Consent to allow all radiographs and medical/surgical/hospitalization records of care received elsewhere prior to and during the study period to be shared with the investigator
10. Willing to maintain current activity and exercise levels throughout the study
11. Willing and able to comply with clinic visits and study-related procedures and willing to provide follow-up information related to any JR surgery that occurs within the period of time covered by their intended participation in the study
12. Able to understand and complete study-related questionnaires

Year 2:

Note: Any Year 1 patient attending their week 52 visit on or after 26 March 2020 will no longer have the option to enroll into Year 2.

1. Completed the treatment period of Year 1
2. Did not permanently discontinue study drug during Year 1
3. Received no less than 10 of the 13 planned doses of SC study drug during the treatment period of Year 1
4. Provide informed consent for Year 2
5. Willing to continue to maintain current activity and exercise levels throughout Year 2

Exclusion Criteria include, but are not limited to, the following:

1. Non-compliance with the Numeric Rating Scale (NRS) recording during the pre-randomization period
2. History or presence at the screening visit of non-OA inflammatory joint disease, Paget's disease of the spine, pelvis or femur, neuropathic disorders, multiple sclerosis, fibromyalgia, tumors or infections of the spinal cord, or renal osteodystrophy
3. History or presence on imaging of arthropathy, neuropathic joint arthropathy, hip or knee dislocation, extensive subchondral cysts, significant bone collapse or bone loss, or pathologic fractures
4. Trauma to the index joint within 3 months prior to the screening visit
5. Signs or symptoms of carpal tunnel syndrome within 6 months of screening
6. Patient is not a candidate for MRI
7. Is scheduled for a JR surgery to be performed during the study period or who would be unwilling or unable to undergo JR surgery if needed
8. History or presence at the screening visit of autonomic or diabetic neuropathy, or other peripheral neuropathy, including reflex sympathetic dystrophy
9. History or diagnosis of chronic autonomic failure syndrome including pure autonomic failure, multiple system atrophy
10. History of naproxen intolerance, or existence of a medical condition that is high risk for naproxen-associated complications
11. Resting heart rate of <50 beats per minute (bpm) or >100 bpm at the screening or randomization visits
12. History or presence of 2nd or 3rd degree heart block, 1st degree heart block with abnormal Complex of Q, R, and S waves on an electrocardiogram (QRS) complex, or bifascicular block by ECG assessment at the screening visit
13. History or presence of orthostatic hypotension at the screening, prerandomization, or randomization visits
14. History of poorly controlled hypertension
15. Use of systemic corticosteroid within 30 days prior to the screening visit. Intra-articular corticosteroids in the index joint within 12 weeks prior to the screening visit, or to any other joint within 30 days prior to the screening visit
16. Exposure to an anti-Nerve growth factor (NGF) antibody prior to the screening visit or known sensitivity or intolerance to anti-NGF antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3307 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2021-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (139):
- United States (58):
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Tucson Orthopaedic Research Center, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - BioSolutions Clinical Research, La Mesa, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Clinical Research, San Marcos, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Jewett Orthopaedic Clinic, Orlando, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Klein & Associates, MD PA, Cumberland, Maryland
  - Klein & Associates, MD, PA, Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Medex Healthcare Research, New York, New York
  - Buffalo Rheumatology and Medicine, PLLC, Orchard Park, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Hickory Family Practice Associates, Hickory, North Carolina
  - Peters Medical Research LLC, High Point, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Hillcrest Clinical Research, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Clinical Research Solutions, Franklin, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Center for Arthritis and Rheumatic Diseases, Chesapeake, Virginia
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
- CCBR Vejle, Vejle, Denmark
- Germany (4):
  - Synexus Clinical Research GmbH, Leipzig, Saxony
  - Synexus Clinical Research GmbH, Berlin
  - Synexus Clinical Research GmbH, Bochum
  - Synexus Clinical Research GmbH, Frankfurt
- Hungary (8):
  - Qualiclinic Kft., Budapest
  - Synexus Magyarorszag Kft, Budapest
  - Synexus Magyarorszag Kft., Debrecen
  - Synexus Magyarorszag Kft., Gyula
  - BKS Research Kft., Hatvan
  - Hevizgyogyfurdo es Szent Andraes ReumaKorhaz, Hévíz
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktato Korhazak Josa Andras Oktatokorhaza Klinikai Kutatasi Osztaly, Nyíregyháza
  - Synexus Magyarorszag Egeszsegugyi Kft., Zalaegerszeg
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Saules Seimos Medicinos Centras, Jsc, Kaunas
  - Republican Panevezys Hospital, Panevezys
  - Center Outpation Clinic, Public Institution, Vilnius
- Poland (14):
  - Synexus Polska Sp. z o.o Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - MCBK Sc lwona Czajkowska Monika Barney, Grodzisk Mazowiecki, Masovian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp. z o.o., Warsaw, Masovian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdynia, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j., Bialystok
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Malopolskie Centrum Kliniczne, Krakow
  - CLINMEDICA RESEARCH OMC, Spolka z Ograniczona Odpowiedzialnoscia Spolka Komandytowa, Skierniewice
  - Etg Zgierz, Zgierz
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp. z o.o. Jednostka 02 - SOMED - Lodzkie Centrum Osteoporozy, Lodz, Łódź Voivodeship
- Romania (2):
  - Clinica Medicala Synexus Ltd., Bucharest
  - SC Policlinica CCBR SRL, Bucharest
- Russia (5):
  - "SBEIHPE ""Kazan State Medical University"" of MHSD of Russia", Kazan', Tatarstan Republic
  - "CDCR ""Healthy Joints"" L.L.C.", Novosibirsk
  - City Out-Patient Clinic #109, Saint Petersburg
  - Samara Regional Clinical Hospital n.a.V.D.Seredavin, Samara
  - "State Autonomous Healthcare Institution of Yaroslavl Oblast ""Clinical Hospital #3""", Yaroslavl
- South Africa (19):
  - Tread Research-Tygerberg Hospital, Parow, Cape Town
  - Welkom Clinical trial Centre, Welkom, Free State
  - Wits Clinical Research, Johannesburg, Gauteng
  - University of Pretoria, Pretoria, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - Synexus SA Stanza Clinical Research Centre, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Soweto Clinical Trials Centre (CTC), Soweto, Johannesburg
  - Synapta Clinical Research Center, Durban, KwaZulu-Natal
  - Enhancing Care, Durban, KwaZulu-Natal
  - Aliwal Shoal Medical Centre, eMkhomazi, KwaZulu-Natal
  - Mzansi Ethical Research Centre Middleburg, Middelburg, Mpumalanga
  - Langeberg Medicross Medical Centre, Kraaifontein, Western Cape
  - Paarl Research Centre, Paarl, Western Cape
  - Synexus Helderberg Clinical Trial Centre, Somerset West, Western Cape
  - TASK Applied Science, Cape Town
  - Mzansi Ethical Research Centre Cape Town, Cape Town
  - Newtown Clinical Research, Johannesburg
- Spain (6):
  - CETA Leganes, Leganés, Madrid
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - MeDiNova Investigacion y Desarrollo, Madrid
  - Centro De Investigacion Clinica En Enfermedades Cronicas - Cicec, Santiago de Compostela
  - Clínica Nuevas Tecnologias en Diabetes y Endocrinologia (NTDE), Seville
  - Hospital Quiron Salud Infanta Luisa, Seville
- Ukraine (6):
  - "Municipal Establishment ""Cherkasy Regional Hospital of Cherkasy Oblast Council""", Cherkasy
  - Kharkiv City Multispecialty Hospital #18, Kharkiv
  - Medical center of Private High Educational Institute Institute of General Practice-Family Medicine, Kyiv
  - "Subsidiary Company ""Medical Research and Practice Center Medbud of the Public Joint Stock ""Holding Company ""Kyivmiskbud""", Kyiv
  - "Kyiv Railway Clinical Hospital No.2 of branch ""Health Center "" of the PJSC ""Ukrainian Railway""", Kyiv
  - Lviv Regional Hospital for veterans of the war and former political prisoners, Lviv
- United Kingdom (12):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Synexus Scotland Clinical Research Centre, Glasgow, Lanarkshire
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - MediNova North London Dedicated Research Centre, Mount Vernon Hospital, Northwood, Middlesex
  - Synexus North East Clinical Research Centre - Hexham General Hospital, Hexham, Northumberland
  - Synexus Midlands Clinical Research Centre, Birmingham, West Midlands
  - Synexus Wales Clinical Research Centre, Cardiff
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Synexus Manchester Clinical Research Centre-Manchester Science Park, Manchester
  - Medinova Research East London Clinical Studies Centre, Romford
  - MeDiNova Research Yorkshire Clinical Studies Centre, Shipley
  - MediNova South London Dedicated Research Centre, Sidcup

REFERENCES:
- [Derived] DiMartino SJ, Cicirello H, Magyar A, Eng S, Ho T, Manvelian G, Patel Y, Pervin K, Trinh N, Fetell M, Braunstein N, Geba GP, Dakin P. A phase III, randomised, double-blind, multi-dose, placebo- and naproxen-controlled study to evaluate the efficacy and safety of fasinumab in patients with pain due to osteoarthritis of the knee or hip. RMD Open. 2026 Jan 16;12(1):e006436. doi: 10.1136/rmdopen-2025-006436. PMID 41545313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9157 participants were screened. Of those, 5850 were screen failures. 3307 participants were randomized into the study.
Groups:
- Placebo: Fasinumab-matching placebo administered by subcutaneous (SC) injection, every 4 weeks (Q4W) and naproxen-matching placebo orally (PO), twice a day (BID)
- Naproxen: Fasinumab-matching placebo SC Q4W and naproxen 500 mg PO, BID
- Fasinumab 1 mg SC Q8W: Fasinumab 1 mg SC Q8W and naproxen-matching placebo, orally, BID
- Fasinumab 1 mg SC Q4W: Fasinumab 1 mg SC Q4W and naproxen-matching placebo, PO, BID
- Fasinumab 3mg Q4W: Fasinumab 3 mg SC Q4W and naproxen-matching placebo PO, BID
- Fasinumab 6mg Q8W: Fasinumab 6 mg SC Q8W and naproxen-matching placebo PO, BID
Period: Overall Study
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3mg Q4W | Fasinumab 6mg Q8W
Started | 354 | 1063 | 551 | 1054 | 145 | 140
As Treated | 352 | 1056 | 554 | 1052 | 145 | 139
Completed | 299 | 919 | 465 | 867 | 102 | 99
Not Completed | 55 | 144 | 86 | 187 | 43 | 41
Not completed — Protocol Violation | 11 | 14 | 6 | 13 | 1 | 0
Not completed — Adverse Event | 5 | 21 | 16 | 35 | 2 | 1
Not completed — Lack of Efficacy | 9 | 13 | 9 | 24 | 4 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 2 | 17 | 15
Not completed — Withdrawal by Subject | 24 | 73 | 44 | 97 | 11 | 10
Not completed — Lost to Follow-up | 3 | 12 | 4 | 7 | 8 | 13
Not completed — Death | 3 | 9 | 7 | 9 | 0 | 0
Not completed — Unknown - Not reported | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W | Fasinumab 3mg Q4W | Fasinumab 6mg Q8W | Total
Number analyzed (Participants) | 354 | 1063 | 551 | 1054 | 145 | 140 | 3307
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 212 | 608 | 300 | 584 | 91 | 81 | 1876
  65 - 84 years | 140 | 449 | 247 | 463 | 53 | 57 | 1409
  85 years and over | 2 | 6 | 4 | 7 | 1 | 2 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 807 | 419 | 793 | 96 | 98 | 2478
  Male | 89 | 256 | 132 | 261 | 49 | 42 | 829
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 26 | 13 | 38 | 6 | 6 | 101
  Not Hispanic or Latino | 339 | 1032 | 537 | 1015 | 139 | 134 | 3196
  Unknown or Not Reported | 3 | 5 | 1 | 1 | 0 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Asian | 11 | 35 | 29 | 37 | 3 | 1 | 116
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 109 | 315 | 166 | 308 | 47 | 47 | 992
  White | 211 | 633 | 307 | 630 | 89 | 86 | 1956
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 23 | 79 | 48 | 79 | 6 | 6 | 241

OUTCOME MEASURES:

1. Primary Outcome: Change in the WOMAC Pain Subscale Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg SC Q4W Compared With That of Participants Treated With Placebo
Description: The WOMAC index is comprised of 24 parameters grouped in 3 subscales (pain-5 questions, physical function -17 questions and stiffness - 2 questions), with 0-10 grading of each question. The scores for each subscale are summed up, divided by number of questions, and each subscale is reported using Numerical Rating Scale score of 0-10. In addition to subscales, a total score is provided as the sum of normalized subscale scores divided by three, and reported using a Numerical Rating Scale score of 0-10. Higher scores indicate worse pain, stiffness and functional limitations.
Time Frame: Baseline to Week 16
Population: Modified Full Analysis Set (mFAS) analysis population; The mFAS excluded additional participants from the Full Analysis Set (FAS) due to regional irregularities noted in some study sites; it was the main analysis population for efficacy endpoints for the fasinumab 1 mg Q4W group. Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 155 | 522
Score on a scale | -1.82 (0.162) | -2.49 (0.098)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Least Squares Mean = -0.68, 95% CI 2-sided [-1.028 to -0.324], Standard Error of Mean 0.180

2. Primary Outcome: Change in the WOMAC Physical Function Subscale Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q4W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: The mFAS excluded additional participants from the Full Analysis Set (FAS) due to regional irregularities noted in some study sites; it was the main analysis population for efficacy endpoints for the fasinumab 1 mg Q4W group. Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 155 | 521
Score on a scale | -1.71 (0.161) | -2.42 (0.096)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg SC Q4W; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean = -0.70, 95% CI 2-sided [-1.046 to -0.346], Standard Error of Mean 0.178

3. Primary Outcome: Change in the WOMAC Pain Subscale Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg SC Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: mFAS Post Protocol Amendment 5 analysis set: For the analysis of fasinumab 1 mg Q8W group comparing to the control groups, only the subset of participants concurrently randomized (ie, after Protocol R475-OA-1611 Amendment 5 Global was implemented) were included. Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 80 | 254
Score on a scale | -2.09 (0.231) | -2.19 (0.144)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg SC Q8W; Test type: Superiority; p = 0.7036, Mixed Models Analysis; Least Squares Mean = -0.10, 95% CI 2-sided [-0.594 to 0.401], Standard Error of Mean 0.254

4. Primary Outcome: Change in the WOMAC Physical Function Subscale Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Fasinumab 1 mg SC Q8W: Fasinumab 1 mg SC Q8W and naproxen-matching placebo, PO, BID
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 80 | 254
Score on a scale | -1.91 (0.223) | -2.09 (0.137)
Statistical Analysis 1: Comparison: Placebo vs Fasinumab 1 mg SC Q8W; Test type: Superiority; p = 0.4605, Mixed Models Analysis; Least Squares Mean = -0.18, 95% CI 2-sided [-0.657 to 0.297], Standard Error of Mean 0.243

5. Secondary Outcome: Change in the Patient Global Assessment (PGA) Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q4W Compared With That of Participants Treated With Placebo
Description: The Patient Global Assessment of OA (PGA) is a patient-rated assessment of current disease state on a 5-point Likert scale (1 = very good; 2 = good; 3 = fair; 4 = poor; and 5 = very poor).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 156 | 526
Score on a scale | -0.64 (0.064) | -0.92 (0.040)

6. Secondary Outcome: Change in the PGA Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q4W Compared With That of Participants Treated With Naproxen
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 492 | 526
Score on a scale | -0.78 (0.040) | -0.92 (0,040)

7. Secondary Outcome: Change In The PGA Scores From Baseline To Week 44 In Participants Treated With Fasinumab 1mg Q4W Compared With That Of Participants Treated With Placebo
Description: as for outcome 5
Time Frame: Baseline to Week 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 123 | 394
Score on a scale | -0.60 (0.074) | -0.79 (0.043)

8. Secondary Outcome: Percentage Of Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Placebo, Who Had A Response At Week 16, With Response Defined As An Improvement By ≥30% In The WOMAC Pain Subscale Scores
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 214 | 639
Percentage of participants | 43.9 | 56.2

9. Secondary Outcome: Percentage of Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Naproxen, Who Had A Response At Week 16, With Response Defined As An Improvement By ≥30% In The WOMAC Pain Subscale Scores
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 644 | 639
Percentage of participants | 50.5 | 56.2

10. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline to Week 16 In Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Naproxen
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 345 | 360
Score on a scale | -2.42 (2.095) | -2.88 (2.099)

11. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline to Week 44 in Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 122 | 391
Score on a scale | -1.69 (0.188) | -2.20 (0.114)

12. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline to Week 44 in Participants Treated With Fasinumab 1 mg Q4W, Compared With That of Participants Treated With Naproxen
Description: as for outcome 1
Time Frame: Baseline to Week 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 381 | 391
Score on a scale | -2.15 (0.115) | -2.20 (0.114)

13. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to the Average Score Across Weeks 4, 8, 12 and 16, in Participants Treated With Fasinumab 1 mg Q4W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 192 | 595
Score on a scale | -1.37 (0.137) | -2.25 (0.088)

14. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to the Average Score Across Weeks 36, 40 and 44 in Participants Treated With Fasinumab 1mg Q4W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 36, 40 and 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 133 | 426
Score on a scale | -1.50 (0.172) | -1.99 (0.113)

15. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Naproxen
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 485 | 521
Score on a scale | -1.98 (0.101) | -2.42 (0.096)

16. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to Week 44 in Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 122 | 390
Score on a scale | -1.60 (0.186) | -2.07 (0.109)

17. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to Week 44 in Participants Treated With Fasinumab 1mg Q4W, Compared With That of Participants Treated With Naproxen
Description: as for outcome 1
Time Frame: Baseline to Week 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 378 | 390
Score on a scale | -2.00 (0.113) | -2.07 (0.109)

18. Secondary Outcome: Change In WOMAC Pain Subscale Scores From Baseline To The Average Score Across Weeks 4, 8, 12 And 16, in Participants Treated With Fasinumab 1mg Q4W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 192 | 596
Score on a scale | -1.46 (0.140) | -2.30 (0.090)

19. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline To The Average Score Across Weeks 36, 40 And 44 In Participants Treated With Fasinumab 1mg Q4W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 36, 40 and 44
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 133 | 427
Score on a scale | -1.57 (0.184) | -2.06 (0.118)

20. Secondary Outcome: Change in the Patient Global Assessment (PGA) Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 80 | 257
Score on a scale | -0.79 (0.094) | -0.77 (0.057)

21. Secondary Outcome: Change in the PGA Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1 mg Q8W Compared With That of Participants Treated With Naproxen
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 245 | 257
Score on a scale | -0.82 (0.057) | -0.77 (0.057)

22. Secondary Outcome: Change In The PGA Scores From Baseline To Week 44 In Participants Treated With Fasinumab 1mg Q8W Compared With That Of Participants Treated With Placebo
Description: as for outcome 5
Time Frame: Baseline to Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 62 | 193
Score on a scale | -0.74 (0.1115) | -0.75 (0.064)

23. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline to Week 16 In Participants Treated With Fasinumab 1mg Q8W, Compared With That of Participants Treated With Naproxen
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 170 | 171
Score on a scale | -2.41 (0.155) | -2.53 (0.154)

24. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline to Week 44 in Participants Treated With Fasinumab 1mg Q8W, Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 62 | 189
Score on a scale | -1.77 (0.276) | -1.99 (0.163)

25. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to the Average Score Across Weeks 4, 8, 12 and 16, in Participants Treated With Fasinumab 1 mg Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 4, 8, 12 and 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 94 | 291
Score on a scale | -1.61 (0.196) | -2.04 (0.127)

26. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to the Average Score Across Weeks 36, 40 and 44 in Participants Treated With Fasinumab 1mg Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 36, 40 and 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 69 | 210
Score on a scale | -1.62 (0.261) | -1.69 (0.166)

27. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to Week 16 in Participants Treated With Fasinumab 1mg Q8W, Compared With That of Participants Treated With Naproxen
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Naproxen | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 241 | 254
Score on a scale | -2.04 (0.140) | -2.09 (0.137)

28. Secondary Outcome: Change in WOMAC Physical Function Subscale Scores From Baseline to Week 44 in Participants Treated With Fasinumab 1mg Q8W, Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 62 | 189
Score on a scale | -1.76 (0.262) | -1.90 (0.157)

29. Secondary Outcome: Change In WOMAC Pain Subscale Scores From Baseline To The Average Score Across Weeks 4, 8, 12 And 16, in Participants Treated With Fasinumab 1mg Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 4, 8, 12 and 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 94 | 291
Score on a scale | -1.73 (0.202) | -2.11 (0.131)

30. Secondary Outcome: Percentage Of Participants Treated With Fasinumab 1mg Q8W, Compared With That of Participants Treated With Placebo, Who Had A Response At Week 16, With Response Defined As An Improvement By ≥30% In The WOMAC Pain Subscale Scores
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 102 | 304
Percentage of participants | 53.9 | 52.3

31. Secondary Outcome: Change in WOMAC Pain Subscale Scores From Baseline To The Average Score Across Weeks 36, 40 And 44 In Participants Treated With Fasinumab 1mg Q8W Compared With That of Participants Treated With Placebo
Description: as for outcome 1
Time Frame: Baseline to average score across weeks 36, 40 and 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fasinumab 1 mg SC Q8W
Number analyzed (Participants) | 69 | 210
Score on a scale | -1.69 (0.271) | -1.80 (0.169)

32. Secondary Outcome: Number of Participants With Adjudicated Arthropathy (AA) (as Confirmed by Adjudication) - Year 1
Time Frame: Baseline to Week 52
Population: The Year 1 safety analysis set (SAF - Year 1) includes all randomized patients from the FAS who received any study drug; it is based on the treatment received (as treated); Here 'n' = Number of evaluable participants at a specified point in time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 352 | 1056 | 554 | 1052
Participants | 4 | 27 | 40 | 102

33. Secondary Outcome: Number of Participants With AA (as Confirmed by Adjudication) - Year 2
Time Frame: First dose of study drug in Year 2 through week 104E
Population: The Year 2 safety analysis set (SAF - Year 2) includes all participants who received at least 1 dose of the Year 2 study drug; it is based on the treatment received during Year 2 (as treated); Here 'n' = Number of evaluable participants at a specified point in time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 137 | 402 | 193 | 371
Participants | 2 | 7 | 11 | 53

34. Secondary Outcome: Number of Participants With AA (as Confirmed by Adjudication) - Year 1 and Year 2
Time Frame: Day 1 through week 104E (Extension)
Population: SAF - Year 2: included all participants who received at least 1 dose of the Year 2 study drug; it was based on the treatment received during Year 2 (as treated). Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 353 | 1056 | 553 | 1052
Participants | 6 | 33 | 50 | 152

35. Secondary Outcome: Number of Participants With Destructive Arthropathy (DA) (as Confirmed by Adjudication) - Year 1
Time Frame: Baseline to Week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 352 | 1056 | 554 | 1052
Participants | 0 | 1 | 2 | 7

36. Secondary Outcome: Number of Participants With DA (as Confirmed by Adjudication) - Year 2
Time Frame: First dose of study drug in Year 2 through week 104E
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 137 | 402 | 193 | 371
Participants | 0 | 0 | 0 | 4

37. Secondary Outcome: Number of Participants With DA (as Confirmed by Adjudication) - Year 1 and Year 2
Time Frame: Day 1 through week 104E
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 353 | 1056 | 553 | 1052
Participants | 0 | 1 | 2 | 11

38. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) - Year 1
Time Frame: Baseline to Week 52
Population: The Year 1 safety analysis set (SAF - Year 1) includes all randomized participants from the FAS who received any study drug; it is based on the treatment received (as treated); Here 'n' = Number of evaluable participants at a specified point in time.
Measure: Number; unit: Events
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 352 | 1056 | 554 | 1052
Events | 1063 | 3641 | 1985 | 3901

39. Secondary Outcome: Number of TEAEs - Year 2
Time Frame: First dose of study drug in Year 2 through week 104E
Population: SAF - Year 2: included all participants who received at least 1 dose of the Year 2 study drug; arm assignment was based on the treatment received during Year 2 (as treated). Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Number; unit: Events
Groups:
- Year 2 Naproxen: Fasinumab-matching placebo SC Q4W and naproxen 500 mg PO, BID; Year 2 naproxen arm contains participants from Year 1 Placebo arm and Year 1 naproxen arm
- Year 2 Fasinumab 1 mg SC Q8W: Fasinumab 1 mg SC Q8W and naproxen-matching placebo, orally, BID
- Year 2 Fasinumab 1 mg SC Q4W: Fasinumab 1 mg SC Q4W and naproxen-matching placebo, PO, BID
Arm/Group | Year 2 Naproxen | Year 2 Fasinumab 1 mg SC Q8W | Year 2 Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 554 | 190 | 385
Events | 973 | 277 | 808

40. Secondary Outcome: Number of TEAEs - Year 1 and Year 2
Time Frame: Day 1 through week 104E
Population: as for outcome 34
Measure: Number; unit: Events
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 353 | 1056 | 553 | 1052
Events | 1317 | 4348 | 2271 | 4712

41. Secondary Outcome: Number of Participants With at Least 1 Sympathetic Nervous System (SNS) Dysfunction Adverse Event of Special Interest (AESI) - Year 1
Time Frame: Baseline to Week 52
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 352 | 1056 | 554 | 1052
Participants | 1 | 0 | 0 | 0

42. Secondary Outcome: Number of Participants With at Least 1 Sympathetic Nervous System (SNS) Dysfunction Adverse Event of Special Interest (AESI) - Year 2
Time Frame: First dose of study drug in Year 2 through week 104E
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Year 2 Naproxen | Year 2 Fasinumab 1 mg SC Q8W | Year 2 Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 554 | 190 | 385
Participants | 0 | 0 | 0

43. Secondary Outcome: Number of Participants With at Least 1 Sympathetic Nervous System (SNS) Dysfunction Adverse Event of Special Interest (AESI) - Year 1 and Year 2
Time Frame: Day 1 through week 104E
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 353 | 1056 | 553 | 1052
Participants | 1 | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With at Least 1 Peripheral Sensory Neuropathy AESI That Require a Neurology or Other Specialty Consultation - Year 1
Time Frame: Baseline to Week 52
Population: Safety Analysis Set (SAF) - Year 1 included participants randomized to fasinumab 1 mg Q4W, fasinumab 1 mg Q8W, naproxen, and placebo. Here 'n' = Number of evaluable participants at the specified point in time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 352 | 1056 | 554 | 1052
Participants | 18 | 43 | 29 | 70

45. Secondary Outcome: Number of Participants With at Least 1 Peripheral Sensory Neuropathy AESI That Require a Neurology or Other Specialty Consultation - Year 2
Time Frame: First dose of study drug in Year 2 through week 104E
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Year 2 Naproxen | Year 2 Fasinumab 1 mg SC Q8W | Year 2 Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 554 | 190 | 385
Participants | 16 | 6 | 12

46. Secondary Outcome: Number of Participants With at Least 1 Peripheral Sensory Neuropathy AESI That Require a Neurology or Other Specialty Consultation - Year 1 and Year 2
Time Frame: Day 1 through week 104E
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 353 | 1056 | 553 | 1052
Participants | 23 | 51 | 35 | 82

47. Secondary Outcome: Number of Participants With Any Type of All-Cause Joint Replacement (JR) in Year 1
Time Frame: Baseline to Week 52
Population: Safety Analysis Set (SAF)-Year 1. For participants with events, number of participant years is calculated up to the date of the first event; for participants without event, it corresponds to the length of the study participation in Year 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 352 | 1056 | 554 | 1052
Participants | 12 | 33 | 31 | 67

48. Secondary Outcome: Number of Participants With Any Type of All-Cause JR in Year 2
Time Frame: First dose of study drug in Year 2 through week 104E
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Year 2 Naproxen | Year 2 Fasinumab 1 mg SC Q8W | Year 2 Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 554 | 190 | 385
Participants | 22 | 12 | 33

49. Secondary Outcome: Number of Participants With Any Type of All-Cause Joint Replacement (JR) - Year 1 and Year 2
Time Frame: Day 1 through week 104E
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen | Fasinumab 1 mg SC Q8W | Fasinumab 1 mg SC Q4W
Number analyzed (Participants) | 353 | 1056 | 553 | 1052
Participants | 19 | 47 | 44 | 100

ADVERSE EVENTS:
Time Frame: From first dose up to week 124
Description: As treated population
Groups:
- Fasinumab 1mg Q8W: Fasinumab 1 mg SC Q8W and naproxen-matching placebo, PO, BID
- Fasinumab 1mg Q4W: Fasinumab 1 mg SC Q4W and naproxen-matching placebo PO, BID
Arm/Group | Placebo | Naproxen | Fasinumab 1mg Q8W | Fasinumab 1mg Q4W | Fasinumab 3mg Q4W | Fasinumab 6mg Q8W
All-Cause Mortality (participants affected / at risk) | 5/352 | 13/1056 | 12/554 | 13/1052 | 0/145 | 0/139
Serious Adverse Events (participants affected / at risk) | 49/352 | 103/1056 | 81/554 | 175/1052 | 7/145 | 6/139
Other Adverse Events (participants affected / at risk) | 215/352 | 687/1056 | 382/554 | 727/1052 | 41/145 | 58/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=352) | Naproxen (N=1056) | Fasinumab 1mg Q8W (N=554) | Fasinumab 1mg Q4W (N=1052) | Fasinumab 3mg Q4W (N=145) | Fasinumab 6mg Q8W (N=139)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (11) | 10 (11) | 8 (9) | 1 (1) | 2 (3)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 13 (13) | 44 (53) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 3 (3) | 6 (6) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer helicobacter (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 7 (7) | 7 (7) | 4 (4) | 17 (20) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 5 (6) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 2 (2) | 3 (3) | 4 (4) | 8 (8) | 0 (0) | 1 (1)
Joint resurfacing surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fistula (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tone disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudodementia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=352) | Naproxen (N=1056) | Fasinumab 1mg Q8W (N=554) | Fasinumab 1mg Q4W (N=1052) | Fasinumab 3mg Q4W (N=145) | Fasinumab 6mg Q8W (N=139)
Arthralgia (Musculoskeletal and connective tissue disorders) | 76 (117) | 232 (357) | 152 (228) | 284 (467) | 13 (16) | 30 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (51) | 117 (160) | 83 (112) | 124 (155) | 4 (5) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (27) | 62 (82) | 34 (41) | 65 (88) | 2 (2) | 3 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 (23) | 34 (41) | 22 (29) | 47 (57) | 1 (1) | 2 (3)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 27 (28) | 38 (45) | 109 (126) | 3 (3) | 8 (8)
Nasopharyngitis (Infections and infestations) | 28 (37) | 92 (122) | 54 (64) | 95 (125) | 5 (5) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 25 (27) | 90 (106) | 41 (51) | 92 (111) | 5 (5) | 6 (6)
Urinary tract infection (Infections and infestations) | 24 (29) | 86 (105) | 41 (45) | 79 (101) | 4 (4) | 5 (5)
Influenza (Infections and infestations) | 24 (30) | 55 (70) | 31 (41) | 70 (85) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 19 (20) | 50 (61) | 30 (34) | 41 (46) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 67 (109) | 216 (548) | 127 (308) | 236 (588) | 13 (21) | 8 (10)
Carpal tunnel syndrome (Nervous system disorders) | 15 (16) | 20 (23) | 26 (32) | 58 (69) | 4 (6) | 5 (5)
Constipation (Gastrointestinal disorders) | 8 (8) | 65 (75) | 12 (12) | 22 (23) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 12 (12) | 54 (72) | 27 (35) | 33 (41) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 31 (34) | 77 (88) | 36 (41) | 55 (59) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT03161093/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03161093/SAP_001.pdf